CLINICAL TRIAL: NCT07310017
Title: The Effects of Yoga Exercises With and Without Virtual Reality on Core Stabilization, Balance, and Stress in University Students
Brief Title: Yoga With and Without VR for Core, Balance, and Stress in University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-38
Record Dates: First submitted 2025-11-26; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Health-Related Behavior
Keywords: Mind-body intervention; Immersive therapy; Breathing exercise; Relaxation
MeSH Terms: conditions — Health Behavior | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Yoga Group (Experimental)
  Interventions: Other: Yoga; Other: Virtual Reality
- Traditional Yoga Group (Active Comparator)
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — A structured yoga program designed to improve core stability, postura balance, and stress management. The traditional yoga sessions will focus on breathing control, static and dynamic postures, and progressive muscles engagements. Each session last 30 minutes it's supervised by a physiotherapist, and takes place in a quiet room to minimise external distractions.
Other: Virtual Reality — The VR environment will be created by the MetaQuest 2 which is a immersive virtual realty headset. During the application, the environment will be chosen by the participants among pre-decided virtual environments, such as forest or ocean. According to the environment, the objects around the participants will move with their sounds. The sounds will be only related to the environment like the bird sound, waterfall sound or the wave sound. There is no instruction in the environment.
  Arms: Virtual Reality Yoga Group

SUMMARY:
The present study aims to investigate the combined and comparative effects of yoga exercise performed with and without virtual reality (VR) support on stress levels, core stabilization, and balance in university students aged 18-30. Participants will be screened using validated stress assessment tools to ensure inclusion of individuals with moderate to high perceived stress. Eligible participants will then be randomly assigned to one of two groups:(1) a virtual reality yoga group (VRYG), in which yoga sessions are delivered through immersive VR environments with therapist-guided breathing and movement instruction; and (2) a Traditional Yoga Group (TYG), in which the same therapist will give the same breathing and movement instructions without VR.

Both groups will undergo 12 supervised sessions over a period of four weeks (three sessions per week, each lasting 30 minutes). The intervention protocol includes a structured series of yoga postures designed to target trunk stability, flexibility, and balance, along with breathing techniques such as diaphragmatic breathing and the 4-7-8 method to promote relaxation and stress reduction. The VR group will perform these exercise within calming, immersive virtual environments,while the control group will perform them in a quite,well-lit physical space.

Outcome measures will be collected at baseline and after completion of the intervention. Psychological stress will be evaluated using the Depression, anxiety, and stress scale (DASS-21) with a focus on the stress sub-scale.Physiological indicators, including heart rate and blood pressure will be recorded at rest. Core stabilization will be assessed through plank and side-plank endurance tests, while balance will be evaluated using both static (single-leg stance) and dynamic (Y-Balance Test) protocols. These measures will allow for a comprehensive analysis of the intervention's effects on both mental and physical domains of health.

ELIGIBILITY:
Inclusion Criteria:

* University student aged 18-30
* Moderate-to-high perceived stress levels (DASS-21)
* No contraindications for yoga or VR use

Exclusion Criteria:

* Diagnosed psychological conditions requiring treatment
* Musculoskeletal limitations that prevent participation
* Use of medications affecting stress
* Current participation in structured stress-reduction programs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Stress level Balance performance(Y-balanced test) | Through study completion, an average of 1 month
  Stress will be measured by the Depression, Anxiety, and Stress Scale (DASS-21) - Stress Subscale
  The DASS-21 Stress Subscale evaluates the participants' perceived stress levels over the past week. It consists of seven items rated on a 4-point scale ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). The stress subscale focuses on symptoms such as difficulty relaxing, nervous tension, irritability, and feeling easily upset.
  Total scores are calculated by summing the item scores and multiplying by two to obtain a standardized value. Higher scores indicate greater stress levels. This assessment was used to determine the changes in stress levels before and after the intervention.
Heart rate | Through study completion, an average of 1 month
  Heart rate (beats per minute/bpm) will be measured to assess the physiological stress response. Measurements will be taken using a digital heart rate monitor while participants are seated comfortably. Each participant rested for five minutes prior to the measurement to ensure accuracy. The heart rate will be recorded three times at one-minute intervals, and the average of the three readings will be used for analysis. A decrease in post-intervention heart rate indicates improved relaxation and reduced physiological stress.
Blood pressure | Through study completion, an average of 1 month
  Systolic and Diastolic blood pressure (in mmHg) will be assessed to evaluate cardiovascular responses associated with stress and relaxation. Measurements will be taken using an automatic digital sphygmomanometer on the participant's dominant arm while seated. Participants rested for at least five minutes before the first reading. Three consecutive readings will be obtained, and the average of the systolic and diastolic values will be calculated for analysis. Lower post-intervention readings reflect improved cardiovascular regulation and reduced stress levels.

SECONDARY OUTCOMES:
Core Stabilization-Plank | Through study completion, an average of 1 month
  Core stability was assessed using the plank and side plank endurance tests, which measure the ability of trunk muscles to maintain a neutral spine position against gravity.
  Plank test: Participants support their body on forearms and toes, maintaining a straight line from head to heels. The duration (second) that the position is held is recorded. The test will be repeated three times with rest intervals, and the mean duration will be used for analysis. Longer holding times indicate better core endurance and stabilization.
Core Stabilization-Side Plank | Through study completion, an average of 1 month
  Core stability was assessed using the plank and side plank endurance tests, which measure the ability of trunk muscles to maintain a neutral spine position against gravity.
  Side plank test: Participants rest on one forearm and the side of one foot while keeping the body aligned. The duration (seconds) maintained on each side is recorded. The test will be repeated three times with rest intervals, and the mean duration will be used for analysis. Longer holding times indicate better core endurance and stabilization.
Static balance | Through study completion, an average of 1 month
  Static balance will be evaluated using the single-leg stance test, which measures postural control and neuromuscular coordination. Participants will stand on one leg without support, arms by their sides, and eyes closed. The time (seconds) until balance is lost or the raised foot touches the ground is recorded.
  Each leg will be tested three times with short rest intervals, and the best time for each leg is used in the analysis. Longer durations indicate superior static balance ability.
Dynamic balance | Through study completion, an average of 1 month
  Dynamic balance will be measured using the Y-Balance Test (YBT), which assesses the participant's ability to maintain postural control while reaching in multiple directions.
  Participants stand barefoot on one leg at the center of a Y-shaped grid and extend the opposite leg in three directions-anterior, posteromedial, and posterolateral-without losing balance.
  The distance reached in each direction is measured in centimeters and normalized to leg length using the following written formula:
  Composite Score Percentage (%) equals the sum of the three reach distances (anterior, posteromedial, and posterolateral) divided by three times the leg length, then multiplied by one hundred.
  Higher composite scores reflect better dynamic balance and neuromuscular control.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Öğr. Üyesi Çiçek Günday, Asst. Prof., Principal Investigator — Istinye University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Fizyoterapi ve Rehabilitasyon Uygulama ve Araștırma Merkezi (İSÜFİZYOTEM), Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No